CLINICAL TRIAL: NCT04440254
Title: Natural History of Cardiac Rhythm and Conduction Disorders in Patients with Fabry Disease Evaluated by Long-Term Implantable Holter ECG
Brief Title: Long Duration Holter ECG in Fabry Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C19-57
Record Dates: First submitted 2020-06-12; First posted 2020-06-19 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — Embryo Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ONE (Other): One single group of patients
  Interventions: Diagnostic Test: Implantation (subcutaneous) of a marketed miniaturized Holter ECG recording device

INTERVENTIONS:
Diagnostic Test: Implantation (subcutaneous) of a marketed miniaturized Holter ECG recording device — Subcutaneously implanted under local anesthesia of the device on the presternal or subclavicular region

SUMMARY:
The main objective is to assess the occurrence of cardiac arrhythmias and conduction disorders during a three-year follow-up using implantable Holter ECG monitoring in 40 patients with Fabry disease. The secondary objectives are to analyze the correlations of these anomalies with changes in cardiac MRI and echocardiographic parameters as biological parameters and overall severity of the disease assessed by MSSI.

DETAILED DESCRIPTION:
The main objective of this non-blinded, monocentric non-randomized study is to assess the occurrence of cardiac arrhythmias and conduction disorders (sinus dysfunction, branch block [BB], atrioventricular block [BAV], sustained [TVS] or non-supported [TVNS] ventricular tachycardias, atrial fibrillation [AF] during a three-year follow-up in 40 patients with Fabry disease (half with left ventricular hypertrophy) using an implantable Holter ECG device (Medtronic Reveal-LINQ™). The secondary objectives are to analyze the correlations (at 1, 2 and 3 years) of these anomalies with the modifications of :

* cardiac MRI [Magnetic Resonance Imaging] data at inclusion [M0] and at 36 months [M36] (left ventricular hypertrophy [HVG], amplitude of the T1 signal, extent of fibrosis); MRIs will be performed before implantation and after removal of the Holter to avoid the reading artifacts linked to the device.
* echocardiographic measurements of the left ventricle (overall longitudinal strain systolic [SGL] and ejection fraction [FE])
* biological parameters (BNP or NT-proBNP, ultra-sensitive troponin and Lyso-Gb3)
* the overall severity of the disease assessed by MSSI (Mainz Severity Score Index), DFG and proteinuria

ELIGIBILITY:
Inclusion Criteria:

* Male patient
* Age greater than or equal to 18 years on the day of inclusion
* Presence of a morbid mutation for MF
* Signature of the informed consent form
* Absence of significant valve disease, verified on medical file (absence stenosis or regurgitation <2+ in color Doppler on a scale 1 to 4+ by extension of the jet)
* No history of known or documented myocardial infarction nor CAD
* No pacemaker or ICD
* no history of AF, NSVT, high-degree AV block
* Correct echogenicity
* No treatment by corticosteroid or immunosuppressive drugs
* creatinine clearance >/= 30 Ml/mn
* LVEF ≥ 50% by ultrasound and / or MRI
* No contraindication to MRI (or claustrophobia) and gadolinium injection
* Affiliation to the French social security insurance

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of cardiac arrhythmias and conduction disorders | 3 years

SECONDARY OUTCOMES:
Correlations between electrical disorders and changes in MRI/ultrasonic data (LV mass, T1 signal, fibrosis extent , systolic strain, ejection fraction), concentrations of BNP, troponin, Lyso-Gb3, MSSI score and renal function | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- 20 Rue Leblanc, HEGP/PARCC, 75015 Paris, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No